CLINICAL TRIAL: NCT05582785
Title: Low Field Magnetic Resonance Imaging Assessment With Outpatients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Sherwin Chan MD PhD, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00002266
Record Dates: First submitted 2022-09-08; First posted 2022-10-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Conditions Requiring a Brain Magnetic Resonance Imaging, Head Computerized Tomography, or Head Ultrasound

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hyperfine (Experimental): For patients that have standard of care head imaging, we will do a secondary analysis to compare their standard of care MRI, CT and/or US exams with Hyperfine MRI exams.
  Interventions: Diagnostic Test: Hyperfine MRI

INTERVENTIONS:
Diagnostic Test: Hyperfine MRI — Patients who have a standard of care MRI, CT or US will undergo a low-field MRI utilizing Hyperfine either at the patient's bedside or in the department of Radiology. Results of the Hyperfine MRI will not be used for clinical care and will only be available to members of the research team for review.

SUMMARY:
The objective of the study is to perform imaging assessments of an early stage magnetic resonance imaging (MRI) system on patients using low field magnetic strength.

ELIGIBILITY:
Inclusion Criteria

Outpatients at CMH Adele Hall Radiology ages 0 days to 22 years are eligible for enrollment.

Exclusion Criteria

No additional sedation will be given as part of this study and that sedation, if already administered, will not be altered for study purposes.

Any patient who has a contraindication to having an MRI, such as:

Non-MRI conditional implanted device or device that is not able to be removed for MRI examination

Ages: 0 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of hyperfine MRI versus conventional MRI, CT and/or US | Through study completion, an average of 3 years
  Sensitivity and specificity of hyperfine MRI versus conventional MRI, CT and/or US

CONTACTS AND LOCATIONS:
Overall Officials: Sherwin Chan, MD PhD, Principal Investigator — Children's Mercy
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No